CLINICAL TRIAL: NCT02940158
Title: The Effect of Various Serving Sizes of Lentils and Other Starchy Meals on Post Prandial Blood Glucose Response and Insulin
Brief Title: Various Serving Sizes of Lentils on Blood Glucose and Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Saskatchewan Pulse Growers (Other)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16AU001
Record Dates: First submitted 2016-09-25; First posted 2016-10-20 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: lentils; diabetes; glycemia; insulin; glucose
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1/2 cup (Other): 1/2 cup serving size arm
  Interventions: Other: 1/2 cup- small red lentil; Other: 1/2 cup- small green lentil; Other: 1/2 cup- corn; Other: 1/2 cup- macaroni; Other: 1/2 cup- white potato; Other: 1/2 cup- white rice
- 1/4 cup (Other): 1/4 cup serving size arm
  Interventions: Other: 1/4 cup- Small red lentil; Other: 1/4 cup- Small green lentil; Other: 1/4 cup- corn; Other: 1/4 cup- macaroni; Other: 1/4 cup- white potato; Other: 1/4 cup- white rice

INTERVENTIONS:
Other: 1/4 cup- Small red lentil
  Arms: 1/4 cup
Other: 1/4 cup- Small green lentil
  Arms: 1/4 cup
Other: 1/4 cup- corn
  Arms: 1/4 cup
Other: 1/4 cup- macaroni
  Arms: 1/4 cup
Other: 1/4 cup- white potato
  Arms: 1/4 cup
Other: 1/4 cup- white rice
  Arms: 1/4 cup
Other: 1/2 cup- small red lentil
  Arms: 1/2 cup
Other: 1/2 cup- small green lentil
  Arms: 1/2 cup
Other: 1/2 cup- corn
  Arms: 1/2 cup
Other: 1/2 cup- macaroni
  Arms: 1/2 cup
Other: 1/2 cup- white potato
  Arms: 1/2 cup
Other: 1/2 cup- white rice
  Arms: 1/2 cup

SUMMARY:
The purpose of this study is to assess the effects of consuming either 1/2 or 1/4 cup servings of lentils on post-prandial blood glucose and insulin as compared to 4 types of starchy foods (corn, macaroni, white potato, white rice).

DETAILED DESCRIPTION:
Eligible participants will undergo a total of 6 study visits. During each visit, a fasted blood sample will be taken by fingerprick, and approximately 500 µL of blood will be dripped into a collection tube. The participant will then consume a meal of either: two types of lentils, corn, macaroni, white rice, or white potato. All study days will be randomized. Each meal will be served in either 1/4 or 1/2 cup servings depending on the study block. Six more blood samples will be taken by fingerprick at 15, 30, 45, 60, 90 and 120 minutes after the beginning of the meal.

ELIGIBILITY:
Inclusion Criteria

* Healthy men and women
* Age 18-40 years
* Body mass index (BMI) 20-30 kg/m2

Exclusion Criteria:

* Tobacco use
* Pregnant or breastfeeding
* Fasting blood glucose ≥ 7.0 mmol/L
* Two hour blood glucose ≥ 11.1 mmol/L after consuming 75g glucose drink (Oral Glucose Tolerance Test beverage)
* Any major medical condition including a history of AIDS or hepatitis
* Medical or surgical event requiring hospitalization within 3 months of randomization
* Any medications except a stable dose (3 months) of oral contraceptives, blood pressure or statin medications
* Blood pressure >140/90 mm Hg
* Natural health products (NHPs) used for glycemic control
* Probiotic supplements
* Dietary fibre supplements
* Consumption of >4 servings of pulses per week
* Food allergy or non-food life threatening allergy
* Shift workers
* Alcohol consumption >14 drinks/week or >4 drinks/sitting
* Recent or intended significant weight loss or gain (>4 kg in previous 3 months)
* Elite athletes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Postprandial Blood Glucose | 2 hours Postprandial
Postprandial Blood Insulin | 2 hours postprandial

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No